CLINICAL TRIAL: NCT05487339
Title: Comparison of Pain Relief and Spread Level in Upper and Lower Lumbar Erector Spinae Plane Block
Brief Title: Comparison of Pain Relief After Upper and Lower Lumbar Erector Spinae Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Keimyung Medical School
Record Dates: First submitted 2022-08-01; First posted 2022-08-04 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Pain, Chronic
Keywords: Pain, Lumbar, Spread
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- upper lumbar ESPB group (Active Comparator): Group where ESPB is performed at L2 with local anesthetic mixture 20 ml
  Interventions: Procedure: Erector spinae plane block
- lower lumbar ESPB group (Active Comparator): Group where ESPB is performed at L4 with local anesthetic mixture 20 ml
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — fascial plane injection guided by fluoroscopy device

SUMMARY:
The primary endpoint of this study was to identify if eretor spinae plane block (ESPB) has any effect in relieving low back pain or leg pain in lumbar radiculopathy. The secondary endpoint was to compare the number of spread level when upper or lower lumbar ESPB was performed.

DETAILED DESCRIPTION:
The erector spinae plane block (ESPB) is a less invasive, safer, and technically easy alternative procedure to conventional neuraxial anesthetic techniques. In contrast to common neuraxial techniques such as paravertebral and epidural injections, the ESPB targets an interfascial plane which is far from the spinal cord, root, and pleura. First applied to thoracic neuropathic pain, currently ESPB is being applied to postoperative pain control and includes variable clinical situations. In the abdomen and thoracic wall, thoracic ESPB can be applied for pain control after cardiac surgery, video-assisted thoracic surgery, laparoscopic cholecystectomy, and thoracotomy. Recently, favorable postoperative pain control after lumbar spinal or lower limb surgeries has been reported with lumbar ESPB. In addition, ESPB has also been used for chronic pain conditions in the upper and lower extremities. To investigate the possible mechanism of action of the ESPB, many previous studies have focused on examining the physical spread of the injected agent. Commonly, contrast dye injections in human cadavers have been utilized to assess the spread level. Physical spread level was determined using various methods including direct dissection or sectioning, computed tomography (CT), thoracoscopic inspection, or magnetic resonance imaging (MRI) with radiocontrast injection. Apart from human cadaver studies, physical spread level has been evaluated in alive patients using a variable volume of local anesthetics mixed with radiocontrast. However, these studies are limited by the small number of included patients. Therefore, the exact spread level of injected local anesthetics remains unclear and a study on a large number of patients is still required

ELIGIBILITY:
Inclusion Criteria:

* lumbar disc herniation
* lumbar foraminal stenosis
* lumbar central stenosis
* lumbar spondylolisthesis
* severe level of spine at L3-4
* numerical rating scale > 4
* back pain functional scale < 45
* duration of pain > 1 month
* patients who can fully understand all items described in BPFS

Exclusion Criteria:

* Allergy to local anesthetics or contrast medium
* Pregnancy
* Spine deformity
* Prior history of lumbar spine surgery
* No previous lumbar MRI or CT
* Patients with coagulation abnormality
* Incorrect level of ESPB

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale changes among 5 times period | baseline, 10 minutes after ESPB, 1 week after ESPB, 2 weeks after ESPB, 4 weeks after ESPB
  numerical rating scale changes after ESPB among 5 times period
back pain function scale changes among 2 times period | baseline, 4 weeks after ESPB
  back pain function scale changes after ESPB among 2 times period

SECONDARY OUTCOMES:
spread level in the cranio-caudal direction | baseline, 1 minute after ESPB
  fluoroscopic contrast medium spread level in the cranio-caudal direction

CONTACTS AND LOCATIONS:
Overall Officials: Ji H Hong, Ph.D, Principal Investigator — Keimyung University
Locations (1):
- Hong ji HEE, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No